CLINICAL TRIAL: NCT04221360
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability After Oral Administration of High Dose CKD-375 and D390 in Healthy Adults.
Brief Title: A Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD-375
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A92_02BE1920
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): * Period 1: D390
  * Period 2: CKD-375
  Interventions: Drug: CKD-375; Drug: D390
- Group 2 (Experimental): * Period 1: CKD-375
  * Period 2: D390
  Interventions: Drug: CKD-375; Drug: D390

INTERVENTIONS:
Drug: CKD-375 — Test drug, QD, PO
Drug: D390 — Reference drug, QD, PO

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety and tolerability of CKD-375.

DETAILED DESCRIPTION:
A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability After Oral Administration of High Dose CKD-375 and D390 in Healthy Adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult who is 19 ~ 55 years at the time of screening
2. Body weight more than 55 kg for male and more than 50kg for female
3. BMI more than 18.5 kg/m2 or less than 27.0 kg/m2
4. Females must be menopause or surgical infertility
5. Males who have consented to the use of appropriate pregnancy contraceptive methods up to 28 days after the last investigational product and not to provide sperm
6. Subjects who voluntarily decided to participate and informed consent based upon understanding on the study.

Exclusion Criteria:

1. Subjects who have a history of clinically significant hepatic, renal, nervous, immune, respiratory, urinary, digestion, endocrine, hemato-oncology, cardiovascular systemic disease or psychosis disorder
2. Subjects who has clinically significant dehydration or is vulnerable to dehydration due to poor oral intake
3. Subjects who underwent intravenous administration of radioactive iodine contrast agents (e.g., intravenous urography, venous cholangiography, angiography, computed tomography using contrast agents, etc.) within 48 hours prior to the first dose of the investigational product
4. Subjects who have a significant urinary tract infection or have such a history
5. Subjects who have genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
6. Subjects who have a history of gastrointestinal disorders (Crohn's disease, ulcerative colitis, etc.) or surgery (except simple appendectomy or hernia surgery) that may affect the absorption of the drug
7. Subjects who have a history of clinically significant hypersensitivity to drugs or additives, including components of the investigational product (empagliflozin, metformin)
8. Subjects who are deemed unsuitable as subjects in the screening test performed within 28 days before the administration of investigational product

   * AST, ALT> UNL(Upper Normal Limit)x1.25
   * Total bilirubin > UNL(Upper Normal Limit)x1.5
   * eGFR (Estimated Glomerular Filtration Rate) <60 mL / min / 1.73m2 using the MDRD (Modification of Diet in Renal Disease) formula
   * Positive immunologic serological tests (hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test, syphilis test)
   * After resting for more than 5 minutes, systolic blood pressure> 150 mmHg or < 90 mmHg, diastolic blood pressure> 100 mmHg or <50 mmHg
9. Subjects who have had a history of drug abuse within one year of screening or have tested positive on urine drug screening test
10. Pregnant or lactating women
11. Subjects who have consistently excessively smoked or consumed caffeine or alcohol (caffeine:> 5 cups / day, alcohol:> 210 g / week, cigarettes:> 10 cigarettes / day) or cannot stop smoking, consuming caffeine and alcohol during hospitalization
12. Subjects who took any of the following drugs except for topical without serious systemic absorption and hormonal contraceptives and are deemed that the administered drug may affect in the study or the safety of the subject by the investigator

    * Ethical-the-counter (ETC) drugs and herbal medicines within 14 days of the first administration of the investigational drug
    * Over-the-counter (OTC) drugs, including health foods and vitamin preparations, within 7 days of the first dose of the investigational product
    * Drugs administered by depot injection or through iomplantation in the human body within 30 days of the first dose of investigational product
13. Subjects who have received the investigational product by participating in other clinical trials (including bioequivalence studies) within 180 days before the first dose of the investigational product (For biological agents, this may be based on a longer period of time, considering the half-life)
14. Subjects who donated whole blood within 60 days before the first dose of the investigational product or donated component blood donation within 30 days
15. Subjects who were deemed to be inappropriate to participate in the study by the investigator judgment

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-01-29 (Estimated); Primary Completion 2020-03-06 (Estimated); Study Completion 2020-06-08 (Estimated)

PRIMARY OUTCOMES:
Cmax of D390 and CKD-375 | 0(predose)~48 hours
  Maximum plasma concentration of D390 and CKD-375
AUClast of D390 and CKD-375 | 0(predose)~48 hours
  Area under the plasma concentration-time curve to last concentration of D390 and CKD-375

SECONDARY OUTCOMES:
AUCinf of D390 and CKD-375 | 0(predose)~48 hours
  Area under the plasma concentration-time curve from zero to infinity concentration of D390 and CKD-375
Tmax of D390 and CKD-375 | 0(predose)~48 hours
  Time to maximum plasma concentration of D390 and CKD-375
t1/2 of D390 and CKD-375 | 0(predose)~48 hours
  Half-life of D390 and CKD-375
Vd/F of D390 and CKD-375 | 0(predose)~48 hours
  Apparent volume of distribution of D390 and CKD-375
CL/F of D390 and CKD-375 | 0(predose)~48 hours
  Apparent clearance of D390 and CKD-375

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, M.D., Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Severance Hospital, Soeul, South Korea